CLINICAL TRIAL: NCT01838356
Title: Intracranial Atherosclerosis and Predictors of Post-CABG Depression
Brief Title: Intracranial Atherosclerosis and Depression After Coronary Artery Bypass Graft
Acronym: NOAHS
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1202009664
Record Dates: First submitted 2013-04-15; First posted 2013-04-24 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Depression; Intracranial Atherosclerosis; Coronary Artery Disease
Keywords: Depression; Vascular depression; Intracranial atherosclerosis; Coronary artery disease; Coronary artery bypass graft; Cognitive impairment
MeSH Terms: conditions — Depression; Intracranial Arteriosclerosis; Coronary Artery Disease; Vascular Depression; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment.

SUMMARY:
The purpose of the study is to examine if blood flow in the brain before coronary artery bypass graft surgery has an effect on depression after surgery.

The main hypothesis of the study states that pre-surgical blood flow in the brain will be an independent risk factor for depression after surgery after adjusting for other risk factors such as gender, pre-CABG depression, social support, medical comorbidity burden, socioeconomic status, and neuroticism.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 years or older
* Will be having CABG surgery at the Yale New Haven Hospital
* Be able to provide informed consent
* Have a household telephone
* A fluent English speaker, and possessing no communication barrier
* Be able to come to the study site or to have the study team come to his/her home.
* Has a family member or partner/ friend who could provide collateral information

Exclusion Criteria:

* Has had previous CABG surgery
* History of dementia diagnosis or cognitive impairment (CDR >/= 1)
* Auditory or visual impairment that would interfere with study procedures
* Active alcohol or substance abuse problem based CAGE-AID (endorsing two or more items)
* History of Bipolar Disorder, Schizophrenia, Schizoaffective Disorder, or any Psychotic Disorder by medical history or self-report.
* Presence of non-cardiovascular conditions likely to be fatal within 1 year

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this study will be drawn from cardiac surgery patients at a university-based hospital who will undergo coronary artery bypass graft (CABG) surgery.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2012-09; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pre-surgical intracranial atherosclerosis as measured by transcranial doppler ultrasound relative to depressive symptoms post-surgically as measured by DISH. | 12 months

SECONDARY OUTCOMES:
Examine neurocognitive function relative to post-CABG depression through a series of neurocognitive tests. | 12 months
  Neurocognitive tests are aimed at evaluating memory, processing speed, and global cognition.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yale University School of Medicine, New Haven, Connecticut
  - The Johns Hopkins University, Baltimore, Maryland

REFERENCES:
- [Derived] Choi JJ, Kukla B, Walsh P, Oldham MA, Lee HB. Functional, cognitive, and cerebrovascular aspects of depression before coronary artery bypass graft surgery: Testing the vascular depression hypothesis. Int J Geriatr Psychiatry. 2023 Sep;38(9):e6000. doi: 10.1002/gps.6000. PMID 37684728
- [Derived] Oldham MA, Hawkins KA, Yuh DD, Dewar ML, Darr UM, Lysyy T, Lee HB. Cognitive and functional status predictors of delirium and delirium severity after coronary artery bypass graft surgery: an interim analysis of the Neuropsychiatric Outcomes After Heart Surgery study. Int Psychogeriatr. 2015 Dec;27(12):1929-38. doi: 10.1017/S1041610215001477. Epub 2015 Oct 2. PMID 26423721